CLINICAL TRIAL: NCT04786145
Title: Cryoneurolysis Outcome on Pain Experience (COPE) in Patients With Low-back Pain - a Single-blinded Randomized Controlled Trial
Brief Title: Cryoneurolysis Outcome on Pain Experience (COPE) in Patients With Low-back Pain
Acronym: COPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COPE
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-01

CONDITIONS: Chronic Low-back Pain; Facet Joint Pain; Degeneration Lumbar Spine; Facet Joint Syndrome; Back Pain Lower Back Chronic
Keywords: low-back pain; cryoneurolysis on lower-back pain; Cryoanalgesia; Cryoneurolysis; Cryoneuroablation; Radiofrequency ablation.
MeSH Terms: conditions — Low Back Pain | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: The study is a single-center, blinded randomized controlled trial with two intervention arms and one placebo arm with allocation ratio of 1:1:1. One group receives one treatment of cryoneurolysis, the second group receives radiofrequency ablation and the third group receives placebo (control group).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Outcomes Assessors, physiotherapists and participants are blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cryoneurolysis (Active Comparator): 40 patients are randomized to receive one treatment of cryoneurolysis on the facet joints of three lumbar level corresponding to their facet joint pain generator
  Interventions: Procedure: Cryoneurolysis
- Radiofrequency ablation (Active Comparator): 40 patients are randomized to receive one treatment of radiofrequency ablation on the facet joints of three lumbar level corresponding to their facet joint pain generator
  Interventions: Procedure: Radiofrequency ablation
- Placebo (Sham Comparator): 40 patients are randomized to receive sham treatment. Subjected to similar procedures as cryoneurolysis and radiofrequency ablation, but without active treatment.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Cryoneurolysis — This is a medical procedure that temporarily blocks nerve conduction along peripheral nerve pathways by freezing it. Small probe is inserted in order to freeze the target nerve, can facilitate complete regeneration of the structure and function of the affected nerve.
  Other Names: cryoanalgesia; cryoneuroablation
  Arms: Cryoneurolysis
Procedure: Radiofrequency ablation — This is a medical procedure that temporarily blocks nerve conduction along peripheral nerve pathways. Small needle with an active heating tip is inserted, to destroy the functionality of the target nerve using heat from radiofrequency energy.
  Arms: Radiofrequency ablation
Procedure: Placebo — No active treatment is given.
  Arms: Placebo

SUMMARY:
This study will provide information on the effectiveness of cryoneurolysis for patients with facet joint pain syndrome, and help to establish whether cryoneurolysis should be implemented in clinical practice for this patient population.

DETAILED DESCRIPTION:
Background: Low-back pain, including facet joint pain, accounts for up to 20 percent of all sick leaves in Denmark; among these are patients with facet joint pain syndrome. A proposed treatment option is cryoneurolysis. This study aims to investigate the effect of cryoneurolysis in lumbar facet joint pain syndrome

Methods: A single-center randomized controlled trial (RCT) is performed including 120 participants with chronic facet joint pain syndrome, referred to the Department of Neurosurgery, Aarhus University Hospital. Eligible patients receive a diagnostic anesthetic block, where a reduction of pain intensity >50 % on a numerical rating scale (NRS) is required to be enrolled. Participants are randomized into three groups to undergo either one treatment of cryoneurolysis, radiofrequency ablation or placebo. Fluoroscopy and sensory stimulation is used to identify the intended target nerve prior to administrating the above-mentioned treatments. All groups receive physiotherapy for 6 weeks, starting 4 weeks after treatment. The primary outcome is a reduction in low-back pain intensity and an impression of change in pain after intervention (Patient Global Impression of Change (PGIC)) at 4 weeks follow-up, prior to physiotherapy. Secondary outcomes are quality of life (EQ-5D, SF-36) and level of function (Oswestry Disability Index), psychological perception of pain (Pain Catastrophizing Scale) and depression status (Major Depression Inventory). Data will be assessed at baseline (T0), randomization (T1), day one (T2), 4 weeks (T3), 3 (T4), 6 (T5) and 12 months

ELIGIBILITY:
Inclusion Criteria:

* Low-back pain from facet joint syndrom (facet joint pain) > 3 months' duration with or without neuropathic pain component.
* Low-back pain on Numeric Rating Scale ≥ 4

Exclusion Criteria:

* Presence of nerve root or spinal canal compression; signs of inflammatory or erosive processes in the spine verified on magnetic resonance imaging (MRI).
* Neurological deficits i.e. symptoms of nerve root compression; tingling, numbness, weakness/ paresis, and reflex loss in the lower extremities.
* Major co-morbidity.
* Anti-thrombotic or anti-platelet treatment which cannot be paused for a week.
* Active malignancies.
* Chronic inflammatory disease.
* Known severe psychiatric disease. Patients with mild and well-treated depression and anxiety are not excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
The effect of the intervention, assessed by Patient Global Impression of Change (PGIC) at 4 weeks follow-up | 4 weeks
  The Patient Global Impression of Change (PGIC) is a 7-point patient self-reporting scale of overall improvement after treatment ranging from 1) very much improved, 2) much improved, 3) minimally improved, 4) no change, 5) minimally worse, 6) much worse, or 7) very much worse

SECONDARY OUTCOMES:
Change in Patient Global Impression of Change (PGIC) at day one, three, six and 12 months follow-up. | 1-12 months
  The Patient Global Impression of Change (PGIC) is a 7-point patient self-reporting scale of overall improvement after treatment ranging from 1) very much improved, 2) much improved, 3) minimally improved, 4) no change, 5) minimally worse, 6) much worse, or 7) very much worse.
Change in the Numeric Rating Scale (NRS-11) from baseline to day one, four weeks, three, six and 12 months follow-up | 1-12 months
  The Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain from 0 no pain to 10 worst pain imaginable.
Change in the Pain Catastrophizing Scale (PCS) at baseline, four weeks, three, six and 12 months follow-up | 1-12 months
  The Pain Catastrophizing Scale (PCS) assesses the extent of catastrophic thinking due to low back pain according to 3 components: rumination, magnification, and helplessness.
  It is a self-report measure, consisting of 13 items scored from 0 to 4, resulting in a total possible score of 52. The higher the score, the more catastrophizing thoughts are present.
Change from baseline to six and 12 months follow-up in the Oswestry Disability Index (ODI). | 1-12 months
  The Owestry Disability Index (ODI) comprises 10 sections with 5 questions in each to measure a patient's permanent functional disability. For each section the scores range of 0 to 5, resulting in a total possible score of 50. If all 10 sections are completed the score is calculated as follows: if 16 (total scored) out of 50 (total possible score) x 100 = 32%. The higher the calculated percentage, the more severe the disability is.
Change from baseline to six and 12 months follow-up in the European Quality of Life - 5 Dimensions (EQ5D) | 1-12 months
  The European Quality of Life - 5 Dimensions (EQ5D) comprises five questions on mobility, self care, pain, usual activities, and psychological status with three possible answers for each item (1=no problem, 2=moderate problem, 3=severe problem. A summary index with a maximum score of 1 can be derived from these five dimensions by conversion with a table of scores. The maximum score of 1 indicates the best health state, in each dimension, where higher scores indicate more severe. In addition, there is a visual analogue scale (VAS) to indicate the general health status with 100 indicating the best health status.
Change from baseline to 12 months follow-up for change in Major Depression Inventory (MDI) and the Short Form (36) Health Survey (SF-36) | 1-12 months
  The Major Depression Inventory (MDI) is a self-reporting measure to assess the presence and severity of a depressive disorder. It consists of 10 questions with a total possible score of 50.
  A score of under 20 indicates no depression and a score of more than 29 indicates severe depression.
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. it consists of 8 scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale. The lower the score the more disability while higher scores indicate the less disability .The maximum score of 100 indicates the best possible health state.

CONTACTS AND LOCATIONS:
Overall Officials: Kaare Meier, MD, Ph.D, Study Director — University of Aarhus; Lone Nikolajsen, M.D, Prof., Study Director — University of Aarhus; Maurits Van Tulder, Prof., Study Director — University of Aarhus; Jens Christian H Sørensen, M.D, Prof., Study Director — University of Aarhus
Locations (1):
- Department of Neurosurgery, Aarhus University Hospital, Aarhus, Central Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sundhedsstyrelsen. Anbefalinger for tværsektorielle forløb for mennesker med kroniske lænderygsmerter. 2017 Pdf;1(1.1):1-38.
- [Background] Binder DS, Nampiaparampil DE. The provocative lumbar facet joint. Curr Rev Musculoskelet Med. 2009 Mar;2(1):15-24. doi: 10.1007/s12178-008-9039-y. Epub 2009 Mar 31. PMID 19468914
- [Background] Trescot AM. Cryoanalgesia in interventional pain management. Pain Physician. 2003 Jul;6(3):345-60. PMID 16880882
- [Background] Freynhagen R, Baron R, Gockel U, Tolle TR. painDETECT: a new screening questionnaire to identify neuropathic components in patients with back pain. Curr Med Res Opin. 2006 Oct;22(10):1911-20. doi: 10.1185/030079906X132488. PMID 17022849
- [Background] Schmidt CO, Schweikert B, Wenig CM, Schmidt U, Gockel U, Freynhagen R, Tolle TR, Baron R, Kohlmann T. Modelling the prevalence and cost of back pain with neuropathic components in the general population. Eur J Pain. 2009 Nov;13(10):1030-5. doi: 10.1016/j.ejpain.2008.12.003. Epub 2009 Feb 6. PMID 19201230
- [Background] Cohen SP, Raja SN. Pathogenesis, diagnosis, and treatment of lumbar zygapophysial (facet) joint pain. Anesthesiology. 2007 Mar;106(3):591-614. doi: 10.1097/00000542-200703000-00024. PMID 17325518
- [Background] Wolter T, Deininger M, Hubbe U, Mohadjer M, Knoeller S. Cryoneurolysis for zygapophyseal joint pain: a retrospective analysis of 117 interventions. Acta Neurochir (Wien). 2011 May;153(5):1011-9. doi: 10.1007/s00701-011-0966-9. Epub 2011 Feb 26. PMID 21359539
- [Background] Birkenmaier C, Veihelmann A, Trouillier H, Hausdorf J, Devens C, Wegener B, Jansson V, von Schulze Pellengahr C. Percutaneous cryodenervation of lumbar facet joints: a prospective clinical trial. Int Orthop. 2007 Aug;31(4):525-30. doi: 10.1007/s00264-006-0208-6. Epub 2006 Aug 23. PMID 16927087
- [Background] Bellini M, Barbieri M. Percutaneous cryoanalgesia in pain management: a case-series. Anaesthesiol Intensive Ther. 2015;47(4):333-5. doi: 10.5603/AIT.2015.0045. PMID 26401741
- [Background] Birkenmaier C, Veihelmann A, Trouillier HH, Hausdorf J, von Schulze Pellengahr C. Medial branch blocks versus pericapsular blocks in selecting patients for percutaneous cryodenervation of lumbar facet joints. Reg Anesth Pain Med. 2007 Jan-Feb;32(1):27-33. doi: 10.1016/j.rapm.2006.08.014. PMID 17196489
- [Background] Maas ET, Ostelo RW, Niemisto L, Jousimaa J, Hurri H, Malmivaara A, van Tulder MW. Radiofrequency denervation for chronic low back pain. Cochrane Database Syst Rev. 2015 Oct 23;2015(10):CD008572. doi: 10.1002/14651858.CD008572.pub2. PMID 26495910
- [Background] Kapural L, Provenzano D, Narouze S. RE: Juch JNS, et al. Effect of Radiofrequency Denervation on Pain Intensity Among Patients With Chronic Low Back Pain: The Mint Randomized Clinical Trials. JAMA 2017;318(1):68-81. Neuromodulation. 2017 Dec;20(8):844. doi: 10.1111/ner.12729. No abstract available. PMID 29220124
- [Background] Lee CH, Chung CK, Kim CH. The efficacy of conventional radiofrequency denervation in patients with chronic low back pain originating from the facet joints: a meta-analysis of randomized controlled trials. Spine J. 2017 Nov;17(11):1770-1780. doi: 10.1016/j.spinee.2017.05.006. Epub 2017 May 30. PMID 28576500
- [Background] Leggett LE, Soril LJ, Lorenzetti DL, Noseworthy T, Steadman R, Tiwana S, Clement F. Radiofrequency ablation for chronic low back pain: a systematic review of randomized controlled trials. Pain Res Manag. 2014 Sep-Oct;19(5):e146-53. doi: 10.1155/2014/834369. Epub 2014 Jul 28. PMID 25068973
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Paulsen RT, Carreon L, Busch F, Isenberg-Jorgensen A. A pilot cohort study of lumbar facet joint denervation in patients with chronic low-back pain. Dan Med J. 2019 Mar;66(3):A5533. PMID 30864544
- [Background] Perrot S, Lanteri-Minet M. Patients' Global Impression of Change in the management of peripheral neuropathic pain: Clinical relevance and correlations in daily practice. Eur J Pain. 2019 Jul;23(6):1117-1128. doi: 10.1002/ejp.1378. Epub 2019 Mar 18. PMID 30793414
- [Background] Correll DJ. The Measurement of Pain: Objectifying the Subjective. Pain Management volume 1, 2007, Pages 197-211
- [Derived] Truong K, Meier K, Ahrens LC, Wichmann TO, Zaer H, Tiroke LH, Arvin S, Bazys M, Duel P, Gudmundsdottir G, Carlsen JG, Nikolajsen L, van Tulder M, Sorensen JCH, Rasmussen MM. Cryoneurolysis versus radiofrequency ablation outcome on pain experience in chronic low back pain (COPE): a single-blinded randomised controlled trial. RMD Open. 2024 May 9;10(2):e004196. doi: 10.1136/rmdopen-2024-004196. PMID 38724261
- [Derived] Truong K, Meier K, Nikolajsen L, van Tulder MW, Sorensen JCH, Rasmussen MM. Cryoneurolysis' outcome on pain experience (COPE) in patients with low-back pain: study protocol for a single-blinded randomized controlled trial. BMC Musculoskelet Disord. 2021 May 19;22(1):458. doi: 10.1186/s12891-021-04320-7. PMID 34011351